CLINICAL TRIAL: NCT02165189
Title: A Phase 2 Open-Label Study in Patients With Recurrent Genotype 1 Hepatitis C Post-Orthotopic Liver Transplant to Explore the Safety And Efficacy of Simeprevir and Sofosbuvir With and Without Ribavirin
Brief Title: An Efficacy and Safety Study of Simeprevir and Sofosbuvir With and Without Ribavirin in Participants With Recurrent Genotype 1 Hepatitis C Post-Orthotopic Liver Transplant
Acronym: GALAXY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104281; TMC435HPC2009 (Other: Janssen Scientific Affairs, LLC)
Record Dates: First submitted 2014-06-10; First posted 2014-06-17 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitits C
Keywords: Simeprevir; Sofosbuvir; Ribavirin; Hepatitits C; Hepatitis C virus ribonucleic acid
MeSH Terms: interventions — Simeprevir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Simeprevir plus Sofosbuvir plus Ribavirin (Arm 1) (Experimental): Participants will be administered simeprevir capsule 150 milligram (mg), sofosbuvir 400 mg tablet, and ribavirin 2 x 200 mg tablets (for participants weighing less than 75 kilogram [kg]) or 3 x 200 mg tablets (for participants weighing more than 75 kg weight), orally once daily up to 12 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir; Drug: Ribavirin
- Simeprevir plus Sofosbuvir (Arm 2) (Experimental): Participants will be administered simeprevir capsule 150 mg and sofosbuvir 400 mg tablet orally once daily up to 12 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir
- Simeprevir plus Sofosbuvir (Arm 3) (Experimental): Participants will be administered simeprevir 150 mg capsule and sofosbuvir 400 mg tablet orally once daily 24 weeks.
  Interventions: Drug: Simeprevir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Simeprevir — Participants will be administered simeprevir capsule 150 mg orally once daily up to 12 weeks.
  Arms: Simeprevir plus Sofosbuvir (Arm 2); Simeprevir plus Sofosbuvir plus Ribavirin (Arm 1)
Drug: Sofosbuvir — Participants will be administered sofosbuvir 400 mg tablet orally once daily up to 12 weeks.
  Arms: Simeprevir plus Sofosbuvir (Arm 2); Simeprevir plus Sofosbuvir plus Ribavirin (Arm 1)
Drug: Ribavirin — Participants will be administered ribavirin 2 x 200 mg tablets (for participants weighing less than 75 kilogram ([kg]) or 3 x 200 mg tablets (for participants weighing more than 75 kg) orally once daily up to 12 weeks.
  Arms: Simeprevir plus Sofosbuvir plus Ribavirin (Arm 1)
Drug: Simeprevir — Participants will be administered simeprevir capsule 150 mg orally once daily up to 24 weeks.
  Arms: Simeprevir plus Sofosbuvir (Arm 3)
Drug: Sofosbuvir — Participants will be administered sofosbuvir 400 mg tablet orally once daily up to 24 weeks.
  Arms: Simeprevir plus Sofosbuvir (Arm 3)

SUMMARY:
The purpose of this study is to evaluate sustained virologic response 12 weeks after the end of treatment (SVR12) following 12 weeks of simeprevir plus sofosbuvir with and without ribavirin (RBV) and 24 weeks of simeprevir plus sofosbuvir without RBV in post orthotopic liver transplant participants with recurrent hepatitis (inflammation of the liver) C virus (HCV) Genotype 1 infection.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter (when more than one hospital or medical school team work on a medical research study), partially randomized (study drug is assigned by chance), and open-label (all people know the identity of the intervention) study to explore the safety and efficacy of simeprevir plus sofosbuvir. The study will consist of a screening period (Screening and Baseline), followed by randomization. First 33 non-cirrhotic participants will be randomly assigned in a ratio of 1:1:1 into 1 of 3 treatment arms, and up to 12 cirrhotic participants will be enrolled and all will be assigned to Arm 3. All participants in treatment Arms 1 and 2 will return for treatment visits at Weeks 1, 2, 4, 8, 12, and post-treatment follow-up visits on Weeks 16 and 24. All participants in treatment Arm 3 will return for treatment visits at Weeks 1, 2, 4, 8, 12, 16, 20, and 24, and post-treatment follow-up visits on Weeks 28 and 36. Participants will receive simeprevir plus sofosbuvir and RBV for a 12-week treatment period in Arm 1, simeprevir plus sofosbuvir without RBV for a 12-week treatment period in Arm 2 and simeprevir plus sofosbuvir for a 24-week treatment period in Arm 3. Efficacy will primarily be evaluated by SVR12. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be infected with Hepatitis C virus (HCV) Genotype 1 (1a or 1b) with Baseline HCV ribonucleic acid (RNA) greater than (>) 10,000 international unit per milliliter (IU/mL). Retesting of HCV RNA to assess eligibility will be allowed once, using an unscheduled visit during the Screening period
* Participant must have had an orthotopic liver transplant greater than or equal to (>=) 6 months to 15 years prior to enrollment
* Participant must have had primary liver transplant
* Participant must be on a stable immunosuppressive regimen for at least 3 months prior to the Screening visit. Immunosuppression regimens may include calcineurin inhibitors (for example, tacrolimus), mammalian target of rapamycin (mTOR) inhibitor, mycophenolate mofetil, prednisone, prednisolone less than or equal to (<=) 5 milligram per day (mg/day), other corticosteroids (except systemic dexamethasone), sirolimus, everolimus, or azathioprine. Stable immunosuppression includes normal adjustment of immunosuppressant dose but excludes changes in immunosuppressant medication and/or treatment of rejection.
* Participant's renal function as measured by the Cockcroft Gault formula must be >30 milliliter per minute (mL/min)

Exclusion Criteria:

* Participants received prior treatment with an investigational or Food and Drug Administration (FDA) approved direct-acting antiviral drug for the treatment of hepatitis C. Prior HCV treatment with interferon or peginterferon with or without ribavirin (RBV) is allowed but must have been completed at least 3 months prior to Screening
* Participants with hepatic decompensation defined by any of the following: 1) Any post-liver transplant clinical signs including ascites, hepatic encephalopathy, and/or evidence of varices with or without variceal bleeding, and 2) Child-Turcotte-Pugh (CTP) score >=7
* Participant has (post-transplant) any underlying serious or life-threatening condition, such as severe uncontrolled cardiopulmonary disease, vascular disease, rheumatologic condition, renal failure, dialysis, ongoing systemic infection, uncontrolled malignancy, or other serious illness that would compromise adherence to medications and ability to comply with all aspects of the study protocol
* Any other active, clinically significant disease or clinically significant findings during the Screening period of medical history, physical examination, laboratory testing, or electrocardiogram (ECG) recording that, in the investigator's opinion, would compromise the participant's safety or could interfere with the participant participating in and completing the study. Retesting of laboratory results that lead to exclusion will be allowed once using an unscheduled visit during the Screening period to assess eligibility
* Participant is a woman who is pregnant, breast-feeding, or planning to become pregnant while enrolled in this study or within 6 months after the last dose of ribavirin (or longer when dictated by local regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response After 12 Weeks of end of Treatment (SVR12) | Week 24 or Week 36
  Participants will be considered to have achieved SVR12 if the hepatitis C virus ribonucleic acid (HCV RNA) is less than (<) 15 international unit per milliliter (IU/mL) (detectable or undetectable) at 12 weeks after the end of treatment. End of treatment is at Week 12 (for Arms 1 and 2) or Week 24 (for Arm 3); therefore, outcome will be measured at Week 24 (for Arms 1 and 2) or Week 36 (for Arm 3).

SECONDARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response After 4 Weeks of end of Treatment (SVR4) | Week 16 (for Arms 1 and 2) and Week 28 (for Arm 3)
  Participants will be considered to have achieved SVR4 if the hepatitis C virus ribonucleic acid (HCV RNA) is <15 IU/mL (detectable or undetectable) at 4 weeks after the end of treatment.
Percentage of Participants With Undetectable Hepatitis C Virus Ribonucleic Acid (HCV-RNA) | Weeks 2, 4, 8 and 12 (for all treatment arms) and Weeks 16 20, and 24 (for Arm 3)
  Plasma HCV RNA will be determined using an in vitro nucleic acid amplification test for the quantification of HCV RNA in human plasma using a sensitive assay (COBAS® AmpliPrep/COBAS® TaqMan® HCV Test v2.0 , lower limit of quantification = limit of detection = 15 IU/mL).
Percentage of Participants With Viral Breakthrough | Baseline up to Week 24 (for Arms 1 and 2) and Baseline up to Week 36 (for Arm 3)
  Viral breakthrough is defined as confirmed greater than (>) 1.0 Log10 increase in HCV RNA from nadir or confirmed HCV RNA >100 IU/mL in participants who had previously achieved HCV RNA <15 IU/mL.
Percentage of Participants With Viral Relapse | Baseline up to Week 24 (for Arms 1 and 2) and Baseline up to Week 36 (for Arm 3)
  Participants will be considered to have viral relapse if they meet the following conditions: 1) HCV RNA <15 IU/mL (undetectable) at the end of treatment; and 2) HCV RNA greater than or equal to (>=) 15 IU/mL during the post-treatment follow-up period.
Change From Baseline in Hepatitis C Symptom and Impact Questionnaire Version 4 (HCV-SIQv4) Score at Week 24 (for Arms 1 and 2) and Week 36 (for Arm 3) | Baseline, Week 24 (for Arms 1 and 2) and Week 36 (for Arm 3)
  The HCV-SIQv4 is a self-administered questionnaire containing 33 items classified as 3 categories of scores: 1) Symptom severity score (sum of responses to 29 questions to assess severity or frequency of symptoms associated with HCV or its treatment; 2) Time missed from work/school (sum of responses to 3 questions regarding the impact of symptoms on work/school attendance); 3) Daily activity score (response to 1 question regarding the impact of symptoms on daily activities). Higher HCV SIQv4 scores indicate worse symptom severity, more time missed from work/school, and more impairment in daily activities, respectively. The total score is the sum of scores of these 3 categories.
Change From Baseline in EuroQol 5 - Dimension (EQ-5D) Questionnaire Score at Weeks 4, 8, 12, 16, 20, 24 (for all treatment arms) and Week 36 (for Arm 3) | Baseline, Weeks 4, 8, 12, 16, 20, 24 (for all treatment arms) and Week 36 (for Arm 3)
  The EQ-5D questionnaire is a brief, generic health-related quality of life assessment (HRQOL) that can also be used to incorporate participant preferences into health economic evaluations. The EQ-5D questionnaire assesses HRQOL in terms of degree of limitation on 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) and as overall health using a "thermometer" visual analog scale with response options ranging from 0 (worst imaginable health) to 100 (best imaginable health). Lower scores indicate worsening. EQ-5D scores include EQ-5D valuation index score (a weighted scoring of the 5 dimension scores with a possible range from 0 to 1), EQ-5D visual analog scale (VAS) is a 20 centimeter (cm) vertical VAS with scores ranging from 0 (worst imaginable health) to 100 (perfect health), and EQ5D descriptive system scores (five scores reflecting each of the 5 EQ-5D health dimensions ranging from 0 [no limitation] to 4 [incapacity]).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Janssen Scientific Affairs, LLC
Locations (11):
- United States (11):
  - Aurora, Colorado
  - Gainesville, Florida
  - Miami, Florida
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - New York, New York
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Dallas, Texas

REFERENCES:
- [Derived] O'Leary JG, Fontana RJ, Brown K, Burton JR Jr, Firpi-Morell R, Muir A, O'Brien C, Rabinovitz M, Reddy R, Ryan R, Shprecher A, Villadiego S, Prabhakar A, Brown RS Jr. Efficacy and safety of simeprevir and sofosbuvir with and without ribavirin in subjects with recurrent genotype 1 hepatitis C postorthotopic liver transplant: the randomized GALAXY study. Transpl Int. 2017 Feb;30(2):196-208. doi: 10.1111/tri.12896. Epub 2017 Jan 20. PMID 27896858
- See also: A Phase 2 Open-label Study in Patients With Recurrent Genotype 1 Hepatitis C Postorthotopic Liver Transplant to Explore the Safety and Efficacy of Simeprevir and Sofosbuvir With and Without Ribavirin. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_7051&studyid=7064&filename=(CR104281)_CSR%20.pdf